CLINICAL TRIAL: NCT00326677
Title: Primary Prevention of Major Depression in Later Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Stephen Thomas, Professor Health Services Administration and Director, Maryland Center for Health Equity, University of Maryland, College Park
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0601117
Record Dates: First submitted 2006-05-15; First posted 2006-05-17 (Estimated); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Depression
Keywords: Depression Prevention; Prevention of Depression; Depression in the Elderly; Late Life Depression; Depression in Old Age; Treatment of Depression in Primary Care Patients; Sub syndromal depression; Minor Depression
MeSH Terms: conditions — Depression | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Problem Solving Therapy — 6 to 8 Problem Solving Therapy sessions over the course of 6 to 16 weeks followed by 3 booster PST sessions over the course of 2 years
Behavioral: Dietary Education — 6 to 8 Diet Education sessions over the course of 6 to 16 weeks followed by 3 booster Diet Education sessions over the course of 2 years

SUMMARY:
The Institute of Medicine has called for studies of "indicated" preventive interventions to reduce the incidence of mental illness in persons already symptomatic but not yet presenting with fully developed clinical syndromes.

The investigators' Advanced Center for Interventions and Services Research in Late Life Mood Disorders has embraced the development and testing of preventive interventions as one of its key objectives. The investigators propose to test the following hypotheses related to primary prevention of major depressive episodes in old age, focusing on elderly patients who have symptoms of emotional distress but who are not yet presenting with the full syndrome of a major depressive episode.

Hypothesis 1: Problem solving therapy (PST) will be superior to an attention-only control (dietary education) in lowering the two-year incidence of episodes of syndromal major depression in already symptomatic elderly primary care patients.

Hypothesis 2: PST will also prevent higher levels of depressive symptoms and associated disabilities, over a two-year period of follow-up.

DETAILED DESCRIPTION:
306 participants will be randomly assigned to either problem solving therapy or to a dietary education control. PST will consist of 6 to 8 sessions, distributed over 6 to 16 weeks, teaching participants a structured process of problem definition, generation of potential solutions, evaluation and choice of solution, and its implementation. The dietary education control will consist of 6 to 8 sessions also, distributed over 6 to 16 weeks. Subjects assigned to the DIET condition will receive education in healthy eating practices (e.g., food pyramid, types of food and calories recommended for people age 60 and above, tips on shopping for healthy food, food preparation, and healthy eating behavior). Subjects will be followed up to 2 years. Length of study is 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or greater
* Center for Epidemiological Studies of Depression Scale (CES-D) score of 11 or higher
* Folstein Mini-Mental State score of 24 or higher
* Not currently receiving antidepressant medication or participating in other mental health treatment

Exclusion Criteria:

* Episode of major depression within the past 12 months
* Episode of alcohol or other substance abuse within the past 12 months
* Life time history of bipolar disorder or other psychotic disorder
* Diagnosis of any neurodegenerative disorder or of dementia (Alzheimer's, vascular, or frontotemporal dementia, etc.)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
BDI, Hamilton, FDI scores, SCID diagnosis of major depression | Over the course of 2 years

SECONDARY OUTCOMES:
CES-D, ISEL,Folstein Mini-Mental, MOS-SF8,BSI, EXIT, Hopkins Verbal Learning Test, PTSD Checklist, Social Problem Solving Inventory, PSQI, CIRS-G, RAND 12 | over the course of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Reynolds III, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Altmann HM, Gebara MA, Albert SM, Morse JQ, Reynolds CF, Thomas SB, Stahl ST. Interpersonal Support Domains Associated With Symptoms of Posttraumatic Stress Among Older Black and White Adults. J Clin Psychiatry. 2023 May 29;84(4):22m14634. doi: 10.4088/JCP.22m14634. PMID 37256634
- [Derived] Kasckow J, Morse J, Begley A, Anderson S, Bensasi S, Thomas S, Quinn SC, Reynolds CF 3rd. Treatment of post traumatic stress disorder symptoms in emotionally distressed individuals. Psychiatry Res. 2014 Dec 15;220(1-2):370-5. doi: 10.1016/j.psychres.2014.06.043. Epub 2014 Jun 28. PMID 25107318
- [Derived] Stahl ST, Albert SM, Dew MA, Lockovich MH, Reynolds CF 3rd. Coaching in healthy dietary practices in at-risk older adults: a case of indicated depression prevention. Am J Psychiatry. 2014 May;171(5):499-505. doi: 10.1176/appi.ajp.2013.13101373. PMID 24788282
- [Derived] Reynolds CF 3rd, Thomas SB, Morse JQ, Anderson SJ, Albert S, Dew MA, Begley A, Karp JF, Gildengers A, Butters MA, Stack JA, Kasckow J, Miller MD, Quinn SC. Early intervention to preempt major depression among older black and white adults. Psychiatr Serv. 2014 Jun 1;65(6):765-73. doi: 10.1176/appi.ps.201300216. PMID 24632760